CLINICAL TRIAL: NCT00673530
Title: Effect of an Evidence Based Clinical Nutrition Concept on Clinical Outcomes in Hospitalized Patients With Malnutrition When Severity of Disease is Taken Into Consideration
Brief Title: Clinical Nutrition Concept for Hospitalized Patients With Malnutrition
Acronym: NUTRICORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Stefan N. Willich, Charité University Medical Center, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUTRICORE
Record Dates: First submitted 2008-05-01; First posted 2008-05-07 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2009-02

CONDITIONS: Malnutrition
Keywords: Hospital malnutrition; Nutritional Status; Nutrition Assessment; Enteral Nutrition; Parenteral Nutrition; Severity of illness index; cost analysis
MeSH Terms: conditions — Malnutrition; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): evidence based clinical nutrition concept
  Interventions: Behavioral: evidence based clinical nutrition concept
- 2 (Other): care as usual
  Interventions: Behavioral: care as usual

INTERVENTIONS:
Behavioral: evidence based clinical nutrition concept — The evidence based nutrition concept comprise a routine malnutrition screening for hospitalized patients, the implementation of an evidence based guideline for clinical nutrition in the participating hospital, education training of the clinical staff and thereby optimal clinical nutrition for malnourished hospitalized patients.
  Other Names: Optimized clinical nutrition concept
  Arms: 1
Behavioral: care as usual — Unchanged treatment of hospital patients without interference by the study.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether there is a positive correlation between an evidence based clinical nutrition concept and relevant clinical outcomes in malnourished hospitalised patients when severity of disease is adjusted.

DETAILED DESCRIPTION:
Patients have been consecutively screened at admission by SGA (Subjective-Global-Assessment)-Score and NRS 2002 (Nutritional-Risk-Screening)-Score in the departments of surgery and internal medicine. The nutrition status of each patient is combined with clinical data, utilization data and direct costs on the basis of clinical homogenous patient clusters. Risk-Adjustment was provided by the Disease-Staging-Scale (MEDSTAT/Thomson Healthcare, Ann Arbor MI), which allows patient classification by diagnosis and co morbidities including age and gender. The risk adjustment scales run by routine data sets from german inpatient G-DRG system. In the control period the effects of usual nutrition care are documented. During the intervention period an implementation of an interdisciplinary evidence-based guideline for screening and clinical nutrition was introduced in each participating hospital.

The issue is to describe the relation between risk-adjusted malnutrition status and clinical outcomes and costs.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* internal or operative admission diagnosis in participating hospitals

Exclusion Criteria:

* Patients with demand for emergency care
* Patients with demand for intensive care
* Patients with hospital day-care
* Patients unwilling to participate or unable to comply with the protocol in the control group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10242 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | At least 3 months each group, 6 months for both groups

SECONDARY OUTCOMES:
all cause hospital mortality | At least 3 months each group, 6 months for both groups
complication rate | At least 3 months each group, 6 months for both groups
hospital readmission rate | 1 Month each group
Economic devices (direct costs of inpatient care and reimbursement) | At least 4 months each group, 7 months for both groups

CONTACTS AND LOCATIONS:
Overall Officials: Stefan N Willich, Prof. Dr., Study Director — Charite University, Berlin, Germany
Locations (4):
- Germany (4):
  - Städtisches Klinikum Ansbach, Ansbach
  - Kliniken Südliche Weinstraße Landau, Bad Bergzaben
  - Evangelische und Johanniter Kliniken, Duisburg
  - Kreiskrankenhaus Hameln, Hamelin